CLINICAL TRIAL: NCT04979104
Title: A Post-market Study Evaluating Clinical and Radiographic Early Outcomes pf Hip Arthroplasty With SL Cementless Stem.
Brief Title: Hip Arthroplasty With SL Cementless
Status: Completed | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-36
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Hip Replacement
Keywords: Cementless femoral stem; Hip arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SL Cementless: Since the trial is not comparative, the only arm implies the use of the investigational device (SL cementless femoral stem)
  Interventions: Procedure: Hip arthroplasty with SL Cementless

INTERVENTIONS:
Procedure: Hip arthroplasty with SL Cementless — Total or partial hip arthroplasty with implant of SL cementless femoral stem.

SUMMARY:
The study aims to evaluate the clinical, radiographical and patient-reported outcomes measurements up 3 years FU and to assess the survivorship of SL Cementless Stem after partial or total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

All patients that underwent to partial or total hip arthroplasty and implanted with SL cementless stem between Jan 2010 and Jan 2020 at Nemocnice Kyjov Hospital (CZ) in accordance with the indication for use of the product and site standard of practice.

Additional Inclusion criteria:

* Availability of patients' immediate post-operative radiograph (baseline) and of a number of follow-up x-rays that the Principal Investigator deems sufficient for an effective radiographic implant evaluation and stability assessment;
* Patient is willing and able to complete additional follow-up evaluations if needed after signing ICF.

Exclusion Criteria:

* Age < 18 years;
* Female patients who are pregnant, nursing, or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Nemocnice Kyjov Hospital (CZ)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Implant radiographic stability | 3 years FU
  Radiographic implant evaluation and stability assessment of the SL Cementless Stem on collected radiographs as per clinical practice during hospitalization and routine visits.

SECONDARY OUTCOMES:
Clinical outcomes | 6 weeks, 3 months, 1 year, 3 years after surgery
  Assessment of the clinical evaluation of the SL Cemetless Stem used in real life settings over a period of 3 years through PROMs if available and medical evaluation
Implant safety profile | 6 weeks, 3 months, 1 year, 3 years after surgery
  Incidence, type and severity of all Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effect (ADEs), Serious Adverse Device Effects (SADEs) at intraoperatively/discharge, 6 weeks, 3 months, 1 year, 3 years after the implant;

CONTACTS AND LOCATIONS:
Locations (1):
- Nemocnice Kyjov Hospital, Kyjov, CZ Republic, Czechia

IPD SHARING:
Plan to Share IPD: No